CLINICAL TRIAL: NCT04741867
Title: Hasan Kalyoncu University Health Sciences Institute
Brief Title: The Effect of Education Based on Roy Adaptation Model for Infertile Individuals on Adaptation and Coping With Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Ayşe Duygu Özbaş, Instructor, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: Hasan Kalyoncu Unıversity
Record Dates: First submitted 2021-01-26; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Health Education
MeSH Terms: conditions — Health Education | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- receiving health education (Experimental)
  Interventions: Other: Education
- Level of compliance (Experimental)
  Interventions: Other: Education
- Coping with stress (Experimental)
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Patients will be educated to determine their level of coping with stress and their adaptation.

SUMMARY:
Psychosocial counseling applied together with infertility treatment programs makes infertile women more resistant to stress, increases the effectiveness of infertility treatments and encourages infertile patients to continue treatment by improving their mental health.

It appears that learning adaptation strategies in infertile couples is concurrent with health promotion. In addition to medical treatments, it is aimed to add training to be given in accordance with the Roy Adaptation model, to adapt to the process and infertility, and to control stress in infertile individuals in the management of the process.

The study was planned to examine the effect of education based on the roy adaptation model for infertile individuals on adaptation and coping with stress.

ELIGIBILITY:
Inclusion Criteria:

* 18-45age difference

Primary infertility

Exclusion Criteria:

- Secondery infertility

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — infertile woman
Enrollment: 61 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Training effectiveness | 3 months
  The education given will increase adaptation to infertility and coping with existing stress.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Duygu Özbaş, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu Üniversitesi, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No